CLINICAL TRIAL: NCT06249555
Title: VOICE-Characterization of Early Response to Vedolizumab and IL-23 Antagonists in Participants With Crohn's Disease Using Patient-Reported Outcome Measures: A Prospective Observational Study
Brief Title: VOICE-Early Response to Vedolizumab and IL-23 Antagonists in Participants With Crohn's Disease: A Prospective Observational Study
Acronym: VOICE
Status: Recruiting | Type: Observational
Sponsor: Alimentiv Inc. (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK01796
Record Dates: First submitted 2024-01-24; First posted 2024-02-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
Keywords: Vedolizumab; Ustekinumab; Patient reported outcome; IL-23 antagonists; Risankizumab
MeSH Terms: conditions — Crohn Disease | interventions — vedolizumab; Ustekinumab; risankizumab; guselkumab; mirikizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vedolizumab: Group one will include participants who will be starting Vedolizumab as part of routine care.
  Dose, frequency and duration are not mandated as part of the study and are determined by the health care provider.
  Interventions: Drug: Vedolizumab (VDZ)
- IL-23 Antagonists: Group two will include participants who will be starting an IL-23 antagonist as part of routine care.
  Dose, frequency and duration are not mandated as part of the study and are determined by the health care provider.
  Interventions: Drug: Ustekinumab (UST); Drug: Risankizumab (RISA); Drug: Guselkumab (GUS); Drug: Mirikizumab (MIR)

INTERVENTIONS:
Drug: Vedolizumab (VDZ) — Participants will receive VDZ as part of routine care.
  Other Names: Entyvio
  Groups: Vedolizumab
Drug: Ustekinumab (UST) — Participants will receive UST as part of routine care.
  Other Names: Stelara
  Groups: IL-23 Antagonists
Drug: Risankizumab (RISA) — Participants will receive RISA as part of routine care.
  Other Names: Skyrizi
  Groups: IL-23 Antagonists
Drug: Guselkumab (GUS) — Participants will receive GUS as part of routine care.
  Other Names: Tremfya
  Groups: IL-23 Antagonists
Drug: Mirikizumab (MIR) — Participants will receive MIR as part of routine care.
  Other Names: Omvoh
  Groups: IL-23 Antagonists

SUMMARY:
The primary aim of this study is to explore the time course of response to Vedolizumab in participants with CD as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference-short form (SF), as well as other PROMIS domain SFs (fatigue, anxiety, depression, sleep disturbance, physical function, and ability to participate in social roles and activities); other PRO measures will also be assessed.

DETAILED DESCRIPTION:
Vedolizumab (VDZ), a monoclonal antibody that selectively targets intestinal T-cell trafficking, is an effective and safe treatment for moderately to severely active Crohn's disease (CD). Recent evidence from open-label, blinded endpoint studies such as VERSIFY and LOVE-CD provide further support for the efficacy of VDZ in achieving clinical, endoscopic, histologic and radiologic disease improvement in CD. Despite these data, VDZ is generally perceived to have a slower onset of action than other biologics, including tumor necrosis factor (TNF) antagonists and the interleukin (IL)-12/23 antagonist, ustekinumab (UST). The IL-23 antagonist risankizumab (RISA) has been more recently approved for treatment of CD and post-hoc analyses of SEQUENCE trial data showed RISA to be superior to UST for inducing clinical remission at Week 24, and thus, RISA may also be considered to have a quicker onset of action than VDZ. This perception largely emanates from the results of the VDZ pivotal for CD (GEMINI 2) where efficacy was assessed at Week 6 after only 2 doses in a largely refractory population. However, in clinical practice VDZ induction consists of 3 doses of VDZ 300 mg administered intravenously at weeks 0, 2 and 6 instead of the 2 doses used in the pivotal trials. In recent clinical trials, induction endpoints for therapeutics in CD are now typically measured at least after Week 12. Accordingly, it is uncertain whether the generally held perception of a relatively slow onset of action for VDZ is accurate. Moreover, it should also be noted that the perception of a slow onset of action has also been conflated to infer that VDZ is a relatively less effective induction therapy in CD than TNF antagonists or UST. Further data to evaluate these issues are needed.

Rapidity of symptom resolution, which is commonly used as a surrogate for speed of onset, is a priority for patients and clinicians. It is therefore important to better understand the kinetics of symptom improvement captured using patient-reported outcomes (PROs) in patients initiating VDZ for treatment of CD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is an adult 18 years of age or older with confirmed CD, as per standard clinical criteria which may include symptoms, endoscopy, histopathology, and imaging.
2. Participant has active CD and has been prescribed as standard of care (SOC) and is planned to start VDZ or IL-23 antagonist therapy (UST, RISA, or GUS or MIR [if approved for the treatment of CD during the recruitment period for this study]) for the first time in accordance with the product label, as determined by the treating physician.
3. Participant has a baseline PROMIS Pain Interference-SF score ≥ 15 (corresponding T-score ≥ 55) (PROMIS Pain Interference-SF 8a [V1.1]).

   a. Score is calculated by adding score (1 to 5) for each of the 8 subcomponents.
4. Participant has completed all SOC biologic work-up assessments (this may include assessment of tuberculosis, chronic infections, Clostridioides difficile infection and vaccination status per local practice).
5. Ability of participant to participate fully in all aspects of this observational study. Full comprehension of consent language and informed consent must be obtained from the participant and documented.

Exclusion Criteria:

1. Participant has CD-related surgery planned or anticipated during the study.
2. Participant has prior exposure to an advanced therapy for the treatment of CD (biologic or small molecule) other than an anti-TNF (i.e., anti-integrin, anti-IL, Janus kinase inhibitors, or sphingosine-1-phosphate receptor 1). Prior failure or intolerance to 2 or more anti-TNF (i.e., infliximab, adalimumab, or certolizumab pegol) therapies in the past 3 years is also cause for exclusion.
3. Participant has an active infection at baseline requiring intravenous systemic antibiotics.

   Note: The treating physician must have completed all appropriate baseline screening tests as per the product label.
4. Participant has evidence of C. difficile toxin or is prescribed treatment for C. difficile infection, or other intestinal bacterial pathogen, ≤ 2 weeks prior to Screening.
5. Participant has chronic non-inflammatory bowel disease pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in US and Canadian participants with CD prescribed VDZ or IL-23 antagonists for the first time. Approximately 300 participants with CD who are initiating first-time treatment with VDZ or UIL-23 antagonists will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess time of onset of biologic therapy in pain interference | Baseline to Week 14
  Time to meaningful clinical improvement in pain interference, defined as a ≥ 2-point decrease in the PROMIS Pain Interference-SF T-score

SECONDARY OUTCOMES:
To assess time of onset of biologic therapy in multiple QOL and functioning domains | Baseline to Weeks 14, 30, and 52
  Time to meaningful clinical improvement for each individual PROMIS domain, defined as a ≥ 2-point change in the direction of improvement in the respective PROMIS domain T-score (Note: A higher PROMIS domain T-score represents more of the concept being measured. For the Ability to Participate in Social Roles and Activities domain an increase in T-score
To assess the efficacy of therapy in inducing a meaningful clinical improvement in pain interference through Week 52 through a reduction in PROMIS - Pain Interference - Short Form Scores. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in fatigue through Week 52 through a reduction in PROMIS - Fatigue - Short Form Scores. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in anxiety through Week 52 through a reduction in PROMIS - Emotional Distress - Anxiety - Short Form Scores. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in depression through Week 52 through a reduction in PROMIS Emotional Distress - Depression - Short Form. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in sleep disturbance through Week 52 through a reduction in PROMIS - Sleep Disturbance - Short Form. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in physical function through Week 52 through a reduction in PROMIS - Physical Function - Short Form. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess the efficacy of therapy in inducing a meaningful clinical improvement in ability to participate in social roles and activities through Week 52 through a reduction in PROMIS - Ability to Participate in Social Roles and Activities - Short Form. | Baseline to Weeks 14, 30, and 52
  Meaningful clinical improvement in each individual PROMIS domain at Weeks 14, 30, and 52
To assess early change in patient-reported symptoms within the PRO-2 through Week 14. | Baseline to Week 14
  Change in PRO-2 (liquid/very soft stool frequency + abdominal pain) from baseline to Week 14.
To assess early change in patient-reported symptoms within the PROMIS - Pain Interference - Short Form through Week 14 | Baseline to Week 14
  Change in PROMIS Pain Interference-SF from baseline to Week 14.
To assess early change in patient-reported symptoms within the PROMIS - Fatigue - Short Form through Week 14 | Baseline to Week 14
  Change in PROMIS Fatigue-SF scores from baseline to Week 14.
To assess early change in patient-reported symptoms within the PROMIS - Anxiety - Short Form through Week 14 | Baseline to Weeks 2, 6 and 14
  Change in PROMIS Anxiety-SF-scores from baseline to Weeks 2, 6, and 14.
To assess early change in patient-reported symptoms within the PROMIS - Depression - Short Form through Week 14 | Baseline to Weeks 2, 6 and 14
  Change in PROMIS Depression- SF-scores from baseline to Weeks 2, 6, and 14.
To assess early change in patient-reported symptoms within the PROMIS - Sleep Disturbance - Short Form through Week 14 | Baseline to Weeks 2, 6 and 14
  Change in PROMIS Sleep Disturbance- SF-scores from baseline to Weeks 2, 6, and 14.
To assess early change in patient-reported symptoms within the PROMIS - Physical Function - Short Form through Week 14 | Baseline to Weeks 2, 6 and 14
  Change in PROMIS Physical Function- SF-scores from baseline to Weeks 2, 6, and 14.
To assess early change in patient-reported symptoms within the PROMIS - Ability to Participate in Social Roles and Activities - Short Form through Week 14 | Baseline to Weeks 2, 6 and 14
  Change in PROMIS Ability to Participate in Social Roles and Activities- SF-scores from baseline to Weeks 2, 6, and 14.
To evaluate the association between the PRO-2 and each PROMIS domain | Baseline to Weeks 14, 30, and 52
  Correlation between PRO-2 scores and each individual PROMIS domain T-score
  • Correlation between change in PRO-2 scores and change in each individual PROMIS domain T-score
To assess the efficacy of therapy in resolving patient-reported symptoms by obtaining PRO-2 clinical remission, defined as a stool frequency score ≤ 3 and abdominal pain score ≤ 1 using unweighted subscores through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  PRO-2 improvement (defined as a stool frequency score defined as a stool frequency score ≤ 3 and abdominal pain score ≤ 1 using unweighted subscores and no worsening of stool frequency and/or abdominal pain scores from baseline )
To assess the efficacy of therapy in resolving patient-reported symptoms by obtaining PRO-2 clinical response, defined as a decrease in the weighted PRO-2 of ≥ 50% from baseline through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  PRO-2 enhanced clinical response defined as a decrease in the weighted PRO-2 of ≥ 50% from baseline through week 52
To assess the efficacy of therapy in resolving fecal urgency defined by a change in UNRS scores from baseline through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  SIBDQ remission (defined as an SIBDQ score ≥ 60) at Weeks 2, 6, 14, 22, 30, 38, 46, and 52
To assess the efficacy of therapy in resolving patient-reported symptoms and improving health related QOL as shown by SIBDQ improvement, defined as ≥ 9-point increase in the SIBDQ from baseline through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  PRO-2 clinical response (defined as a decrease in the weighted PRO-2 of ≥ 50% from baseline) at Weeks 2, 6, 14, 22, 30, 38, 46, and 52
To assess the efficacy of therapy in resolving patient-reported symptoms and improving health related QOL as shown by obtaining SIBDQ remission, defined as an SIBDQ score ≥ 60 through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  PRO-2 clinical remission (defined as a stool frequency score ≤ 3 and abdominal pain score ≤ 1 using unweighted subscores) at Weeks 2, 6, 14, 22, 30, 38, 46, and 52
To assess the durability of symptom improvement | Baseline to Week 14
  PRO-2 clinical remission at Week 52 among participants who had PRO-2 clinical remission at Week 14
To assess the efficacy of therapy in resolving patient-reported symptoms by obtaining PRO-2 clinical response through week 52. | Baseline to Weeks 2, 6, 14, 22, 30, 38, 46, and 52
  PRO-2 clinical response defined as ≥ 30% decrease from baseline in unweighted stool frequency score or a ≥ 30% decrease from baseline in unweighted abdominal pain scores, with neither increasing from baseline

CONTACTS AND LOCATIONS:
Locations (23):
- United States (10):
  - GI Alliance - Sun City, Sun City, Arizona
  - Digestive and Liver Center of Florida, Kissimmee, Florida
  - Northwestern University, Evanston, Illinois
  - University of Iowa, Iowa City, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of North Carolina, Chapel Hill, North Carolina
  - OR Clinic - East - GI, Portland, Oregon
  - GI Alliance Research Fort Worth, Fort Worth, Texas
  - GI Alliance Research Mansfield, Mansfield, Texas
  - GI Alliance - Bellevue - Washington Gastroenterology, Bellevue, Washington
- Canada (13):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - GNRR Digestive Clinics and Research Center, Brampton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Alimentiv, London, Ontario
  - West GTA Research Inc., Mississauga, Ontario
  - Rajbir Rai Medicine Professional Corporation, Oakville, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Scarborough Center for Inflammatory Bowel Disease, Scarborough Village, Ontario
  - Toronto Immune & Digestive Health Institute Inc., Toronto, Ontario
  - McMaster University Medical Center, Hamilton, Ontatrio
  - Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No